CLINICAL TRIAL: NCT02875444
Title: Measurement of Maximum Diameter of Native Abdominal Aortic Aneurysm by Angio-computed Tomography
Brief Title: Measurement of Maximum Diameter of Native Abdominal Aortic Aneurysm by Angio-CT
Acronym: AAA-angioCT
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2015Ao001
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- group "abdominal aortic aneurysm": Patients with non-operated abdominal aortic aneurysm with angio-CT realized between 01/01 2010 au 04/15/2012
  Interventions: Other: Angio-CT

INTERVENTIONS:
Other: Angio-CT

SUMMARY:
Screening for an abdominal aortic aneurysm, monitoring its growth and evaluation of its risk of rupture are based on the measure of its maximum diameter. The abdominal aortic aneurysm's treatment to prevent its rupture is recommended from a threshold of 50-55 mm in men and of 45-50 mm in women.

The importance of this measure for patient management justify a specific and homogeneous protocol of measure. However, the diversity of methods of measuring the maximum diameter with scanner and ultrasound was shown.

The impact of various angio-CT based measures of maximum AAA diameter, and the impact of reproducibility limits on the decision to operate have never been investigated.

DETAILED DESCRIPTION:
The aims of the study were :

Analyze the consequences on clinical decisions of this wide choice of methodologies for measurement of abdominal aortic aneurysm maximum diameter when using angio-CT; Identify the method of measurement that yields the best agreement for patient management.

ELIGIBILITY:
Inclusion Criteria:

* patients with abdominal aortic aneurysm

Exclusion Criteria:

* inflammatory aneurysm
* false aneurysm
* aneurysm after open repair or stent graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with non-opered abdominal aortic aneurysm with angio-CT realized between 01/01 2010 au 04/15/2012
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum diameter of abdominal aortic aneurysm | Day 0
  Maximum abdominal aortic aneurysm measured using 11 measurement methods

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France